CLINICAL TRIAL: NCT02859727
Title: An Open-label, Non-randomized Extension Study to Evaluate the Long Term Safety, Tolerability, Efficacy and Pharmacokinetics of CDZ173 in Patients with APDS/PASLI (Activated Phosphoinositide 3-kinase Delta Syndrome/p110δ-activating Mutation Causing Senescent T Cells, Lymphadenopathy and Immunodeficiency)
Brief Title: Extension to the Study of Efficacy of CDZ173 in Patients with APDS/PASLI
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: All participant have transitioned to commercial product or compassionate use.
Sponsor: Pharming Technologies B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCDZ173X2201E1; 2016-000468-41 (EudraCT Number)
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Activated PI3Kdelta Syndrome (APDS); PASLI Disease
Keywords: APDS; PASLI; PI3Kdelta; p110delta-activating mutation causing senescent T cells, lymphadenopathy and immunodeficiency; Activated PI3Kdelta Syndrome;
MeSH Terms: conditions — Activated PI3K-delta Syndrome; Lymphadenopathy; Immunologic Deficiency Syndromes | interventions — leniolisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CDZ173 (Experimental): 140mg/day
  Interventions: Drug: CDZ173

INTERVENTIONS:
Drug: CDZ173 — 140 mg/day

SUMMARY:
This study is designed to provide long-term CDZ173 treatment, a selective PI3Kδ inhibitor, to the patients with genetically activated PI3Kδ, i.e., patients with APDS/PASLI who participated in the CCDZ173X2201 study or who were treated previously with PI3Kδ inhibitors other than CDZ173. The study is open-label designed to establish the long-term safety, tolerability, efficay and pharmacokinetics of CDZ173 in the target population.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Paients must have participated in the study CCDZ173X2201 or were treated previously with PI3Kδ inhibitors other than CDZ173.
* Patients who are deemed by the Investigator to benefit from PI3Kδ inhibitor therapy.
* Patients or their legal representatives (for patients under the age of 18 years) must be able to communicate well with the Investigator, to understand and comply with the requirements of the study.
* Documented APDS/PASLI-associated genetic PI3K delta mutation.

Exclusion Criteria:

- Any medically significant disease or condition that is unrelated to APDS/PASLI

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the long term safety and tolerability of CDZ173 in patients with APDS/PASLI | 6 years 3 months
  All safety parameters (including AEs, physical exam, vital signs, ECG, safety laboratory (hematology, blood chemistry, urinalysis))

SECONDARY OUTCOMES:
To evaluate the long term efficacy of CDZ173 to modify health-related quality of life in patients with APDS/PASLI | 6 years
  SF-36 (Short Form 36) Survey and WPAI-CIQ (Work Productivity Activity Impairment plus Classroom Impairment Questionnaire), Visual analogue scales for Physician's Global Assessment (PGA) and Patient's Global Assessment (PtGA), patient narratives by Investigator
To evaluate the long term efficacy of CDZ173 by means of biomarkers reflecting the efficacy of CDZ173 to reduce systemic inflammatory components of the disease in patients with APDS/PASLI | 8 months
  High sensitivity C-reactive protein (CRP), lactate dehydrogenase (LDH), frequencies of infections and other disease complication
To characterize the pharmacokinetics (trough concentration) of CDZ173 in patients with APDS/PASLI | 9 months
  Steady-state trough concentration of CDZ173
• To evaluate the pharmacokinetics and relative bioavailability of CDZ173 film-coated tablets compared to CDZ173 hard-gelatin capsules | up to 6 months
  PK parameters (including but not limited to AUC0-12,ss and Cmax,ss)

CONTACTS AND LOCATIONS:
Locations (8):
- Pharming Investigative Site, Bethesda, Maryland, United States
- Pharming Investigative Site, Minsk, Belarus
- Pharming Investigative Site, Prague, CZE, Czechia
- Pharming Investigative Site, Dresden, Germany
- Italy (2):
  - Pharming Investigative Site, Brescia, BS
  - Pharming Investigative Site, Palermo, PA
- Pharming Investigative Site, Rotterdam, Netherlands
- Pharming Investigative Site, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Rao VK, Kulm E, Grossman J, Buchbinder D, Chong H, Bradt J, Webster S, Sediva A, Dalm VA, Uzel G. Long-term treatment with selective PI3Kdelta inhibitor leniolisib in adults with activated PI3Kdelta syndrome. Blood Adv. 2024 Jun 25;8(12):3092-3108. doi: 10.1182/bloodadvances.2023011000. PMID 38593221
- [Derived] Rao VK, Kulm E, Sediva A, Plebani A, Schuetz C, Shcherbina A, Dalm VA, Trizzino A, Zharankova Y, Webster S, Orpia A, Korholz J, Lougaris V, Rodina Y, Radford K, Bradt J, Relan A, Holland SM, Lenardo MJ, Uzel G. Interim analysis: Open-label extension study of leniolisib for patients with APDS. J Allergy Clin Immunol. 2024 Jan;153(1):265-274.e9. doi: 10.1016/j.jaci.2023.09.032. Epub 2023 Oct 4. PMID 37797893